CLINICAL TRIAL: NCT02630589
Title: Implantation of an Auditory Brainstem Implant for the Treatment of Incapacitating Unilateral Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Principal Investigator, Minke van den Berge, prof. P. van Dijk, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI for tinnitus
Record Dates: First submitted 2015-12-03; First posted 2015-12-15 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Tinnitus
Keywords: tinnitus; auditory brainstem implant; electrical stimulation
MeSH Terms: conditions — Tinnitus | interventions — Auditory Brain Stem Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI implantation (Experimental): All 10 patients included in the study will be neurosurgically implanted with the ABI. This is open label, not blinded. The implant is permanent, but can be switched off.
  Interventions: Device: Auditory brainstem implant

INTERVENTIONS:
Device: Auditory brainstem implant — The ABI will be implanted by the neurosurgeon. The implant is fixed in a bed drilled in the parietal-temporal cortex, and the ABI electrode array is inserted into the lateral recess of the fourth ventricle and placed on the cochlear nucleus. Access to the cochlear nucleus will be made via retrosigmoid transcranial approach.
  Other Names: ABI

SUMMARY:
Tinnitus is the perception of sound or noise in the absence of an external physical source. It is a highly prevalent condition and for a high percentage of patients, there is no satisfying treatment modality. For some people, tinnitus has a very severe impact on quality of life, leading to incapacity for work and sometimes even suicidality. The auditory brainstem implant (ABI) is an implant indicated for the restoration of hearing in patients with an hypo-, or aplasia of the cochlear nerve or with dysfunction of the nerve caused by tumor growth in neurofibromatosis type II. It has been shown that the standard intended effect of an ABI has reduction of tinnitus as a welcome side effect in about 66% of the cases. This is in analogy with the promising effect of a cochlear implant (CI) as a treatment for patients with unilateral tinnitus. In this study, the effect of an ABI on severely invalidating, unilateral, intractable tinnitus will be investigated. The ABI may have an advantage over the CI as tinnitus treatment, because CI-implantation leads to destruction of inner ear structures, leading to profound deafness, while an ABI is presumed to not damage anatomical structures. This is the first study to implant an ABI for the primary aim of tinnitus reduction in an intervention pilot study. In total 10 patients with unilateral, intractable tinnitus and severe hearing loss in the ipsilateral ear, will be implanted with the ABI.

DETAILED DESCRIPTION:
Rationale: Tinnitus is the perception of sound or noise in the absence of an external physical source. It is a highly prevalent condition and for a high percentage of patients, there is no satisfying treatment modality. For some people, tinnitus has a very severe impact on quality of life, leading to incapacity for work and sometimes even suicidality. The auditory brainstem implant (ABI) is an implant indicated for the restoration of hearing in patients with an hypo-, or aplasia of the cochlear nerve or with dysfunction of the nerve caused by tumor growth in neurofibromatosis type II. It has been shown that the standard intended effect of an ABI has reduction of tinnitus as a welcome side effect in about 66% of the cases. This is in analogy with the promising effect of a cochlear implant (CI) as a treatment for patients with unilateral tinnitus. In this study, the effect of an ABI on severely invalidating, unilateral, intractable tinnitus will be investigated. The ABI may have an advantage over the CI as tinnitus treatment, because CI-implantation leads to destruction of inner ear structures, leading to profound deafness, while an ABI is presumed to not damage anatomical structures. This is the first study to implant an ABI for the primary aim of tinnitus reduction.

Objective. To evaluate the efficacy of an ABI for the suppression of unilateral, intractable tinnitus and to establish the safety of the ABI for this new indication.

Study design. This is a single center, non-randomized, prospective cohort, intervention pilot study. There is no control group. In this study, 10 patients will be implanted with an ABI.

Study population. Adult patients with invalidating, unilateral, intractable tinnitus and ipsilateral severe hearing loss are included in this study. All study participants have no significant comorbidity and are mentally competent.

Intervention. All study participants receive an ABI, which will be neurosurgically implanted. The ABI will be switched on 6 weeks after implantation. The surgery and post-surgery follow-up and switch-on procedures are consistent with the intended use of the ABI.

Main study parameters. The primary outcome is change in the Tinnitus Functioning Index (TFI). The endpoint is set at 1 year after implantation. Follow up will take place until 5 years after implantation.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness. The implantation, activation and fitting of the ABI will be performed exactly as described in the existing protocols for intended use, however in this study, the ABI is placed for another indication. Implantation of the ABI requires hospital admission for estimated 4 days. After dismissal, patients visit the outpatient clinic at least 8 times in the first year, depending on the amount of fitting session necessary. Implantation of the ABI is an invasive procedure, which potentially can cause severe complications (meningitis 3,8%, transient hydrocephalus 1,3%, cerebellar contusion 1,2%). Other complication that may occur are infection, bleeding, hearing loss and other cranial nerve dysfunctions. By an extensive training program for the neurosurgeon and presence of the experienced surgeon during the first surgical procedures, the investigators feel that neurosurgical risks and risk of device failure due to inadequate implantation can be limited. In this pilot study, the effects on hearing and tinnitus are still uncertain, however based on the results published in literature the investigators are confident that the effects on both will be positive. Nonauditory side-effects and disappointing results on hearing and/or tinnitus can be well managed by altering stimulation strategy or if necessary, by turning off the device. Tinnitus can be severely invalidating with a large impact on quality of life and the ABI is promising in reducing tinnitus in these patients. This study imposes a significant risk on the study participants. However, the investigators feel that the risks outweighs the potential to ameliorate severely debilitating tinnitus.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral tinnitus
* Severely invalidating tinnitus
* Men or women, age >18yr
* Tinnitus that is present >1 years and was stable during the last year
* Tinnitus that is nonresponsive to indicated conventional existing treatments (hearing aids and cognitive behavioral therapy (CBT)). If a psychologist has indicated that CBT may ameliorate tinnitus complaints, the patient should have tried CBT for long enough time to reasonably argue that these treatments were not successful. This is the same for hearing aids.
* Ipsilateral ear: pure tone audiometry (PTA) thresholds >40dB and <90dB (mean over 1-2-4kHz)
* Functional hearing in the contralateral ear with pure tone audiometry thresholds <35dB (mean over 1-2-4 kHz) and with a minimum Δ25dB compared to the ipsilateral ear.
* Informed consent after extensive oral and written information about the surgery, complications and the uncertain effect of the ABI on tinnitus

Exclusion Criteria:

* Detectable cause for tinnitus that requires causal therapy (e.g. vestibular schwannoma, glomus tumor, otosclerosis, arteriovenous malformation) as investigated by radiological and otological examination
* Psychiatric pathology and/or an unstable psychological situation as declared by a psychiatrist
* Unrealistic expectations as declared by the investigator and/or psychiatrist
* Life expectancy <5 years
* History of blood coagulation pathology
* ASA >II
* Pregnancy
* Anatomic abnormalities that would prevent appropriate placement of the stimulator housing in the bone of the skull
* Anatomical abnormalities or surgical complications that might prevent placement of the Auditory Brainstem Implant Active Electrode Array
* Known intolerance to the materials used in the implant (medical grade silicone, platinum, iridium and parylene C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-07; Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Functioning Index (TFI) | pre-op, 3 months, 6 months, 1, 2,3,4,5 year postoperative
  Unit of measure: Items on a scale.
  The TFI (tinnitus functioning index) is a questionnaire validated to detect changes in tinnitus outcome after an intervention

SECONDARY OUTCOMES:
Pure tone audiometry | pre-op, 3 months, 6 months, 1, 2,3,4,5 year postoperative
  Unit of measure: Fletchers Index (mean of dB on 1-2-4 kHz on pure tone audiometry)
  Change in hearing as a result of ABI implantation is measured by pure tone audiometry and speech audiometry
Tinnitus Handicap Inventory (THI) | pre-op, 3 months, 6 months, 1, 2,3,4,5 year postoperative
  Unit of measure: items on a scale
  This validated questionnaire measures the effect of tinnitus on quality of life of the patient.
Vestibular test | pre-op, 3 months postoperative
  Unit of measure: description of vestibular function ("afunctional", "normal functioning"
  To establish an preoperative situation of both vestibular organs, a standard vestibular testing will be performed.
Visual Analogue Score (VAS) | pre-op, 3 months, 6 months, 1, 2,3,4,5 year postoperative
  Unit of measure: items on a scale.
  The VAS (Visual analog scale) is a subjective measurement scale. Registration of VAS-scores gives the ability to quickly measure the aspects of the tinnitus complaints. It consists of a 100mm-horizontal line with 2 endpoints labeled as 0 and 10. The patient states on a scale from 0-10 how much patient is bothered by the complaint. The VAS-tinnitus annoyance (VAS-TA) was labeled as 0 (not annoyed by tinnitus) and 10 (worst possible annoyed by tinnitus). The VAS-tinnitus loudness (VAS-TL) was labeled as 0 (no tinnitus) and 100 (loudest tinnitus ever).(31). Also, the VAS-scores are measured at every follow up moment in 'on' and 'off' mode of the ABI (which will be blinded for the patient), with estimated 10 minutes between the measurements.
Hospital anxiety and depression scale (HADS) | pre-op, 3 months, 6 months, 1, 2,3,4,5 year postoperative
  Unit of measure: items on a scale.
  The HADS (hospital anxiety and depression scale) is validated in Dutch consists of 14 items, each using a Likert scale (0-3), with subscales for anxiety (seven items) and depression (seven items).(30) The suggested cut-off score (with ranges of 0-21 for each subscale) for screening for possible cases is 8, and for probable cases of anxiety and depression 11. Time to complete the HADS is approximately 10-15.
Tinnitus analysis | pre-op, 3 months, 6 months, 1, 2,3,4,5 year postoperative
  tinnitus tone matching in contralateral ear
ABI-related outcomes | at every change in ABI setting (minimum: switch on, 6 wk after switch on, 3 months, 6 months, 1, 2,3,4,5 year postoperative
  Percentage of time that the ABI was used per day (%), logged days (%).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van den Berge MJC, van Dijk JMC, Metzemaekers JDM, Maat B, Free RH, van Dijk P. An auditory brainstem implant for treatment of unilateral tinnitus: protocol for an interventional pilot study. BMJ Open. 2019 Jun 14;9(6):e026185. doi: 10.1136/bmjopen-2018-026185. PMID 31201186